CLINICAL TRIAL: NCT01715493
Title: Pharmacological Effect of Lysozyme for Chronic Obstructive Pulmonary Disease and Asthma With Sputum Symptom: a Randomised Placebo-controlled Study
Brief Title: Pharmacological Effect of Lysozyme for Chronic Obstructive Pulmonary Disease and Asthma With Sputum Symptom
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LYS-0003
Record Dates: First submitted 2012-09-10; First posted 2012-10-29 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma
Keywords: COPD; Asthma; Lysozyme Hydrochloride
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Muramidase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lysozyme 90 mg (Experimental)
  Interventions: Drug: lysozyme 90 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lysozyme 90 mg — Lysozyme 90 mg three times daily for 4 weeks followed by placebo for 4 weeks (plus usual COPD medication)
  Other Names: PRT10T
  Arms: Lysozyme 90 mg
Drug: Placebo — Lysozyme Matching Placebo three times daily for 4 weeks followed by Lysozyme 90 mg three times daily for 4 weeks (plus usual COPD medication)
  Other Names: PRT10T
  Arms: Placebo

SUMMARY:
The aim of this study was to assess the effectiveness for small airway inflammation of 4 weeks lysozyme administration in Chronic Obstructive Pulmonary Disease (COPD) and/or asthma.

ELIGIBILITY:
Inclusion criteria:

For COPD:

* Over 20 years of age and below 85 years of age
* Smoking history
* Brinkman index 200 or more
* Diagnosis of COPD
* Forced expiratory volume in 1 second (FEV1) of <80% of the predicted value
* Ratio of FEV1 to forced vital capacity (FVC) of <70%
* symptom of expectorated sputum

For Asthma

* Over 20 years of age and below 85 years of age
* Scored between 20 to 24 by ACT (Asthma Control Test)
* Symptom of expectorated sputum
* Diagnosed partly controlled by global initiative for asthma

Exclusion criteria:

* Egg allergy
* Domiciliary oxygen therapy
* Pneumonia or pulmonary tuberculosis
* Patients with severe cardiovascular disorder, severe kidney disorder, severe hepatic disorder, severe hematological disorder
* Cancer

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change of several inflammatory or biochemical marker concentration in inducted sputum | 8 weeks (2 periods each lasting 4 weeks)
Peripheral airway resistance and reactance measured by Impulse oscillometry system, and NO concentration. | 8 weeks (2 periods each lasting 4 weeks)

SECONDARY OUTCOMES:
Monthly reduction in forced expiratory volume in 1 Second (FEV1) | 8 weeks (2 periods each lasting 4 weeks)
Quality of life assessed by CAT (COPD Assessment Test) and ACT (Asthma Control Test) | 8 weeks (2 periods each lasting 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Shibata, Study Director — Drug Fostering and Evoluation Coordination Department, Corporate Regulatory Compliance, Safety and Quality Assurance Headquaters
Locations (1):
- Mizunami, Gifu, Japan